CLINICAL TRIAL: NCT03852498
Title: A Phase 3 Study of Lenti-D Drug Product After Myeloablative Conditioning Using Busulfan and Fludarabine in Subjects ≤17 Years of Age With Cerebral Adrenoleukodystrophy (CALD)
Brief Title: A Clinical Study to Assess the Efficacy and Safety of Gene Therapy for the Treatment of Cerebral Adrenoleukodystrophy (CALD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALD-104; 2018-001145-14 (EudraCT Number)
Record Dates: First submitted 2019-02-13; First posted 2019-02-25 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Adrenoleukodystrophy (CALD)
Keywords: Adrenoleukodystrophy; X-linked adrenoleukodystrophy; Gene therapy; Hematopoietic stem cell
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenti-D Drug Product (Experimental): Participants received a single intravenous (IV) infusion of eli-cel (also referred to as Lenti-D Drug Product) on Day 1 at a dose of > or = 5.0*10^6 CD34+ cells/kilogram (kg). All participants received myeloablative conditioning with busulfan and fludarabine over a number of days prior to drug product infusion.
  Interventions: Genetic: Lenti-D

INTERVENTIONS:
Genetic: Lenti-D — Participants received a single IV infusion of Lenti-D Drug Product.
  Other Names: elivaldogene autotemcel; eli-cel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Lenti-D Drug Product (also known as elivaldogene autotemcel or Skysona, hereafter referred to as eli-cel) after myeloablative conditioning with busulfan and fludarabine in participants with CALD. A participant's blood stem cells will be collected and modified (transduced) using the Lenti-D lentiviral vector encoding human adrenoleukodystrophy protein. After modification (transduction) with the Lenti-D lentiviral vector, the cells will be transplanted back into the participant following myeloablative conditioning. Enrollment and treatment in Study ALD-104 have been completed and further enrollment in this study is not expected, although participants follow-up remains ongoing in the long-term follow-up Study LTF-304 (NCT02698579).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is obtained from a competent custodial parent or guardian with legal capacity to execute a local Institutional Review Board (IRB)/independent ethics committee (IEC) approved consent. Informed assent will be sought from capable participants, in accordance with the directive of the IRB/IEC and with local requirements.
2. Males aged 17 years and younger, at the time of parental/guardian consent and, where appropriate, participant assent.
3. Active CALD as defined by:

   1. Elevated very long chain fatty acids (VLCFA) values, and
   2. Active central nervous system (CNS) disease established by central radiographic review of brain MRI demonstrating: i) Loes score between 0.5 and 9 (inclusive) on the 34-point scale, and ii) Gadolinium enhancement (GdE) on MRI of demyelinating lesions.
4. NFS < or = 1.

Exclusion Criteria:

1. Prior receipt of an allogeneic transplant or gene therapy.
2. Use of statins, Lorenzo's Oil, or dietary regimens used to lower VLCFA levels. Note: participants must discontinue use of these medications at time of consent.
3. Receipt of an investigational study drug or procedure within 3 months before Screening that might confound study outcomes. Use of investigational study drugs is prohibited throughout the course of the study.
4. Any conditions that make it impossible to perform MRI studies (including allergies to anesthetics or contrast agents).
5. Hematological compromise as evidenced by:

   1. Peripheral blood absolute neutrophil count (ANC) count <1500 cells/ cubic millimeter (mm^3), and either
   2. Platelet count <100,000 cells/mm^3, or
   3. Hemoglobin <10 gram per deciliter (g/dL).
6. Hepatic compromise as evidenced by:

   1. Aspartate transaminase (AST) value greater than (>) 2.5 × upper limit of normal (ULN)
   2. Alanine transaminase (ALT) value >2.5 × ULN
   3. Total bilirubin value >3.0 milligram per deciliter (mg/dL), except if there is a diagnosis of Gilbert's Syndrome and the participant is otherwise stable
7. Baseline estimated glomerular filtration rate <70 milliliter per minute (mL/min)/1.73 square meter (m^2).
8. Cardiac compromise as evidenced by left ventricular ejection fraction <40 percent (%).
9. Immediate family member with a known or suspected Familial Cancer Syndrome.
10. Clinically significant uncontrolled, active bacterial, viral, fungal, parasitic, or prion associated infection.
11. Positive for human immunodeficiency virus type 1 or 2 (HIV-1, HIV-2); hepatitis B virus (HBV); hepatitis C virus (HCV); human T lymphotrophic virus 1 (HTLV-1). (Note that participants who have been vaccinated against HBV [positive for HBV surface antibodies] who are negative for other markers of prior HBV infection [e.g., negative for HBV core Ab] are eligible. Participants with past exposure to HBV [hepatitis B core antibody [HBcAb] -positive and/or hepatitis B e-antigen antibody [HBeAb]-positive] are also eligible for the study provided they have a negative test for HBV DNA. Also note that participants who are positive for anti-hepatitis C Ab are eligible as long as they have a negative hepatitis C viral load).
12. Any clinically significant cardiovascular, hematological, or pulmonary disease, or other disease or condition that would be contraindicated for any of the other study procedures.
13. Absence of adequate contraception for fertile participants.
14. Any contraindications to the use of Granulocyte colony-stimulating factor (G-CSF) or plerixafor during the mobilization of HSCs, and any contraindications to the use of busulfan or fludarabine, including known hypersensitivity to the active substances or to any of the excipients in their formulations.
15. Known hypersensitivity to protamine sulfate.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himal Lal Thakar, MD, Study Director — bluebird bio, Inc.
Locations (8):
- United States (3):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Boston Children's Hospital/Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
- Hôpital Robert Debré, Paris, France
- Universitätsklinikum Leipzig AöR, Leipzig, Germany
- Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Prinses Maxima Center, Utrecht, Netherlands
- UCL-ICH/Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency. Appropriately de-identified patient-level datasets and supporting documents may be shared following attainment of applicable marketing approvals associated with this study and consistent with criteria established by bluebird bio and/or industry best practices in order to maintain the privacy of study participants. For enquiries, please contact bluebird bio at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Duncan CN, Bledsoe JR, Grzywacz B, Beckman A, Bonner M, Eichler FS, Kuhl JS, Harris MH, Slauson S, Colvin RA, Prasad VK, Downey GF, Pierciey FJ, Kinney MA, Foos M, Lodaya A, Floro N, Parsons G, Dietz AC, Gupta AO, Orchard PJ, Thakar HL, Williams DA. Hematologic Cancer after Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2024 Oct 10;391(14):1287-1301. doi: 10.1056/NEJMoa2405541. PMID 39383458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 study centers in France, Italy, Germany, the Netherlands, United Kingdom, and United States of America from 24 January 2019 to 24 July 2023.
Pre-assignment Details: A total of 35 male participants were enrolled. All underwent mobilization and were treated with Lenti-D Drug Product also referred to as eli-cel (elivaldogene autotemcel) in this study. For study ALD-104 the Transplant Population (TP), Neutrophil Engraftment Population (NEP), and Intent-to-Treat Population (ITT) are identical.
Groups:
- Lenti-D Drug Product: Participants received a single intravenous (IV) infusion of eli-cel (also referred to as Lenti-D Drug Product) on Day 1 at a dose of greater than or equal to (>=) 5.0 x 10^6 CD34+ cells/kilogram (kg). All participants received myeloablative conditioning with busulfan and fludarabine over a number of days prior to drug product infusion.
Period: Overall Study
Arm/Group | Lenti-D Drug Product
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Transplant Population (TP) consisted of participants who received Lenti-D Drug Product infusion.
Groups:
- Lenti-D Drug Product: Participants received a single IV infusion of eli-cel (also referred to as Lenti-D Drug Product) on Day 1 at a dose of >=5.0 x 10^6 CD34+ cells/kg. All participants received myeloablative conditioning with busulfan and fludarabine over a number of days prior to drug product infusion.
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Alive and Have None of the 6 Major Functional Disabilities (MFDs) at Month 24
Description: The MFDs consisted of loss of communication, cortical blindness, tube feeding, total incontinence, wheelchair dependence, complete loss of voluntary movement. Month-24 MFD-Free survival criteria defined as: alive at 24 months post infusion; have not developed any of the MFDs by 24 months post infusion; have not received rescue cell administration or allo-hematopoietic stem cell transplantation (HSCT) by 24 months post infusion; and have not withdrawn from the study or have not been lost to follow-up by 24 months post infusion.
Time Frame: At Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as participants who have been followed for 24 months (i.e. Rel Day of last contact >=730) or have completed the Month 24 Visit, or discontinued from the study but would have been followed for 24 months if still on the study (i.e. Rel Day of data cut >=730), at the time of the data cut.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 85.7 [69.7 to 95.2]

2. Primary Outcome: Percentage of Participants Who Achieved Neutrophil Engraftment After Drug Product Infusion
Description: Neutrophil engraftment is defined as achieving 3 consecutive absolute neutrophil count (ANC) laboratory values of >= 0.5x10^9 cells/liter (L) (after initial post-infusion nadir) obtained on different days by 42 days postinfusion of eli-cel (Rel Day 43).
Time Frame: By 42 days post-drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants for NE if they achieved neutrophil engraftment by Rel Day 43, or had discontinued or were lost to follow-up before Rel Day 43 without achieving NE, or had been followed to at least Rel Day 43 but had not achieved NE. Participants who discontinued or were lost to follow-up before Rel Day 43 without achieving NE were considered failures for NE.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 100.0 [90.0 to 100.0]

3. Secondary Outcome: Percentage of Participants Without Gadolinium Enhancement (i.e. GdE-) on Magnetic Resonance Imaging (MRI) at Month 24
Description: Percentage of participants without Gadolinium Enhancement (i.e. GdE-) on MRI at Month 24 were reported.
Time Frame: At Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as participants who have completed the Month 24 GdE assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 94.3 [80.8 to 99.3]

4. Secondary Outcome: Number of Participants With Change in Neurologic Function Score (NFS) From Baseline to Month 24
Description: NFS was a 25-point score used to evaluate the severity of gross neurologic dysfunction in cerebral adrenoleukodystrophy (CALD) by scoring 15 symptoms (functional domains) across 6 categories. Listed here are the 15 symptoms followed by their maximal score out of 25 points: a) Hearing/auditory processing problems-1, b) Aphasia/apraxia-1, c) Loss of communication-3, d) Vision impairment/field cut-1, e) Cortical blindness- 2, f) Swallowing/other central nervous system (CNS) dysfunctions-2, g) Tube feeding-2, h) Running difficulties/hyperreflexia-1, i) Walking difficulties/spasticity/spastic gait (no assistance)-1, j) Spastic gait (needs assistance)-2, k) Wheelchair dependence-2, l) Complete loss of voluntary movement-3, m) Episodes of incontinence -1, n) Total incontinence-2, o) Nonfebrile seizures-1. A score of "0"= absence of clinical signs of cerebral disease.
Time Frame: Baseline up to Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as participants who have non-missing Baseline and have completed the Month 24 NFS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Participants
  Change at Month 24: Increased <=3 | 4
  Change at Month 24: Increased > 3 | 2

5. Secondary Outcome: Number of Participants Who Achieved Stable NFS at Month 24
Description: Stable NFS was defined as maintaining an NFS <=4 without an increase of >3 from Baseline. Number of participants who achieved stable NFS at Month 24 were reported.
Time Frame: At Month 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Participants | 33

6. Secondary Outcome: Major Functional Disability (MFD)-Free Survival Rate
Description: MFD-free survival rate was defined as percentage of participants from drug product infusion to either second transplant, MFD, or death due to any cause, whichever occurs first. MFD-free survival rate was analyzed using Kaplan-Meier Analysis. Kaplan-Meier estimated MFD-free survival rate at 24 months after Lenti-D drug infusion was reported.
Time Frame: At 24 months after Lenti-D drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Deaths, MFDs, and rescue cell administration or allo-HSCT are considered events. If a participant did not experience any event, he was to be censored at the Date of Last Contact.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 88.6 [72.4 to 95.5]

7. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate was defined as percentage of participants alive from date of Lenti-D drug product infusion (Day 1) to date of death of all causes. Overall survival rate was censored at the date of last visit if the subject were alive. Participants who are alive were censored at the date of last contact. Overall survival rate was analyzed using Kaplan-Meier Analysis.
Time Frame: At 24 months after Lenti-D drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 100.0 [100.0 to 100.0]

8. Secondary Outcome: Median Detectable Vector Copy Number (VCN) in Peripheral Blood Cells by Month 6
Description: Presence of vector sequences in the genome of cells derived from the originally transduced HSC indicates the presence of transduced cells amongst the HSC precursors. The presence of vector sequences was evaluated throughout the study in whole blood, in selected subpopulations of blood cells (including CD14+ cells), and in bone marrow when indicated. The presence of vector sequences in the genomic DNA of cells was detected using quantitative polymerase chain reaction (qPCR), and results were expressed as vector copy number (VCN; vector copies per diploid genome, c/dg).
Time Frame: By Month 6 post-transplant
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: copies per diploid genome (c/dg)
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 33
copies per diploid genome (c/dg) | 1.05 [0.03 to 3.13]

9. Secondary Outcome: Time to Neutrophil Engraftment (NE) After Drug Product Infusion
Description: Neutrophil engraftment is defined as achieving 3 consecutive absolute neutrophil count (ANC) laboratory values of >= 0.5 x 10^9 cells/liter (L) (after initial post-infusion nadir) obtained on different days by 42 days post-infusion of eli-cel (Rel Day 43). Time to neutrophil engraftment after drug product infusion was reported.
Time Frame: By 42 days post-drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Days | 14.0 [12 to 31]

10. Secondary Outcome: Percentage of Participants With Platelet Engraftment by Month 24
Description: Platelet engraftment was defined as achieving 3 consecutive unsupported platelet counts of >=20 x 10^9 cells/L (after initial post-infusion nadir) obtained on different days while no platelet transfusions were administered for 7 days immediately preceding and during the evaluation period. The first Day of 3 consecutive platelet counts >=20 x 10^9 cells/L was considered the Day of platelet engraftment.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Participants are evaluable for platelet engraftment if they achieved PE by Month 24, or have been followed for at least 24 months if no platelet engraftment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 100.0 [90.0 to 100.0]

11. Secondary Outcome: Time to Platelet Engraftment Post-drug Product Infusion
Description: Platelet Engraftment was defined as achieving 3 consecutive unsupported platelet counts of > or =20 x 10^9 cells/L (after initial post-infusion nadir) obtained on different days while no platelet transfusions were administered for 7 days immediately preceding and during the evaluation period. The first day of 3 consecutive platelet counts >=20 x 10^9 cells/L was the day of PE. Time to platelet engraftment post-drug product infusion by Month 24 was reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Days | 29.0 [14 to 108]

12. Secondary Outcome: Percentage of Participants With Loss of Neutrophil Engraftment Post-drug Product Infusion by Month 24
Description: Participants were considered to have primary engraftment failure if they did not achieve NE by Relative Day 43. A participant was considered to have secondary engraftment failure if they achieved and then subsequently lost NE by the Month 24, i.e., if they met both the conditions; Achieved NE by Relative Day 43 as defined above and had sustained decline in ANC to < 0.5 x 10^9 cells/L for 3 consecutive measurements on different days after Relative Day 43, without alternate etiology. First day of the 3 consecutive ANC decline to < 0.5 x 10^9 cells/L was considered the day of secondary engraftment failure. Percentage of participants with both primary or secondary loss of neutrophil engraftment at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants include participants who, had either primary engraftment failure or secondary engraftment failure by Month 24, or have been followed for at least 24 months if no events.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 0 [0.0 to 10.0]

13. Secondary Outcome: Percentage of Participants Who Underwent a Subsequent Allo- Hematopoietic Stem Cell Transplantation (HSCT) Infusion by Month 24
Description: Percentage of participants who have undergone a subsequent allo-HSCT infusion by Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as those who received subsequent allo-HSCT, or participants who have been followed for at least 24 months (Rel Day of last contact >= 730 or completed Month 24 visit) if no events. Three participants had Subsequent allo-HSCT by Month 24.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 8.6 [1.8 to 23.1]

14. Secondary Outcome: Percentage of Participants Who Experienced Either Acute (>= Grade 2) or Chronic Graft Versus Host Disease (GVHD) at Month 24
Description: Acute GVHD graded on the Acute GVHD Grading Scale (1-4): Grade 1 is characterized as mild disease, Grade 2 as moderate, Grade 3 as severe (involvement of any organ system), and Grade 4 as life-threatening; chronic GVHD was determined by the Investigator. GVHD was seen after an eli-cel participant received a subsequent allogeneic hematopoietic stem cell transplant. No GVHD was seen in participants who did not receive allogeneic stem cell transplants. Grade 2 non-serious GVHD was reported in a participant who received allogeneic transplant post eli-cel infusion. Percentage of participants who experienced either acute (>= Grade 2) or chronic GVHD at Month 24 were reported.
Time Frame: At Month 24
Population: TP consisted of participants who received Lenti- D Drug Product infusion. Evaluable participants are defined as those who have either experienced the event by Month 24 (Rel Day 730) or have been followed for at least 12 months (Rel Day of last contact >= 365) if no events yet.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 2.9 [0.1 to 14.9]

15. Secondary Outcome: Percentage of Participants Who Experienced >= Grade 2 Acute Graft Versus Host Disease (GVHD) by Month 24
Description: Acute GVHD graded on the Acute GVHD Grading Scale (1-4): Grade 1 is characterized as mild disease, Grade 2 as moderate, Grade 3 as severe (involvement of any organ system), and Grade 4 as life-threatening; Acute GVHD was determined by the Investigator. GVHD was seen after an eli-cel participant received a subsequent allogeneic hematopoietic stem cell transplant. No GVHD was seen in participants who did not receive allogeneic stem cell transplants. Grade 2 non-serious GVHD was reported in a participant who received allogeneic transplant post eli-cel infusion. Percentage of participants who experienced >= Grade 2 Acute GVHD at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as those who had >= Grade 2 acute GVHD by Month 24 (Rel Day 730), or have been followed for at least 12 months (Rel Day of last contact >= 365) if no events yet. The case of GVHD was experienced by a participant after receiving allo-HSCT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 2.9 [0.1 to 14.9]

16. Secondary Outcome: Percentage of Participants Who Experienced Chronic GVHD by Month 24
Description: Chronic GVHD graded on the Chronic GVHD Grading Scale as limited or extensive. Chronic GVHD was determined by the Investigator. No chronic GVHD was observed in any participants. Acute GVHD was seen after an eli-cel participant received a subsequent allogeneic hematopoietic stem cell transplant. No GVHD was seen in participants who did not receive allogeneic stem cell transplants. Grade 2 non-serious GVHD was reported in a participant who received allogeneic transplant post eli-cel infusion. Percentage of participants who experienced chronic GVHD by Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants are defined as those who had chronic GVHD by Month 24 (Rel Day 730), or have been followed for at least 12 months (Rel Day of last contact >= 365) if no events yet.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants | 0 [0.0 to 10.0]

17. Secondary Outcome: Percentage of Participants Who Experienced Transplant-related Mortality Through 100 and 365 Days Post-drug Product Infusion
Description: Transplant-related mortality was determined by the investigator and summarized for the following intervals: from Rel Day 1 through 100 days post-drug product infusion (Rel Day 101) and from Rel Day 1 through 365 days post-drug product infusion (Rel Day 366). Percentage of participants who experienced transplant-related mortality through 100 and 365 days post-drug product infusion were reported.
Time Frame: From time of drug product infusion through 100 and 365 days post-drug product infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants include participants who have died from transplant-related causes by Rel Day 101 or 366 respectively or have been followed to at least Rel Day 101 or 366 respectively if no events yet.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants
  Transplant related mortality within 100 days | 0 [0.0 to 10.0]
  Transplant related mortality within 365 days | 0 [0.0 to 10.0]

18. Secondary Outcome: Percentage of Participants With Clinical >= Grade 3 Adverse Events (AEs), All Investigational Medicinal Product-related AEs, All Serious Adverse Events (SAEs), and >= Grade 3 Infections
Description: Adverse event was defined as any untoward medical occurrence associated with the use of a drug product in participants, whether or not considered drug related. SAE was any AE, occurring at any dose and regardless of causality, that resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or was considered an important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent an outcome listed previously. Percentage of participants with clinical >= Grade 3 AEs, all investigational medicinal product-related AEs, all serious adverse events (SAEs), and >= Grade 3 infections were reported.
Time Frame: From date of informed consent up to Month 24
Population: Intent-to-treat (ITT) population consisted of participants who initiated any study procedures, beginning with mobilization by granulocyte colony stimulating factor (G-CSF).
Measure: Number; unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants
  Participants with at least 1 >= Grade 3 AE | 100.0
  Participants with at least 1 AE related to Eli-cel | 20.0
  Participants with at least 1 SAE | 62.9
  Participants with >= Grade 3 infections | 28.6

19. Secondary Outcome: Number of Participants With >= Grade 3 Prolonged Cytopenia on or After Rel Day 60 And Rel Day 100
Description: Number of participants with >= Grade 3 prolonged cytopenia (i.e., decreased platelet counts, decreased neutrophil counts, and/or decreased hemoglobin counts) on or after Rel Day 60 and Rel Day 100 were reported.
Time Frame: Prolonged cytopenias occurring on or after Rel Day 60 and Rel Day 100 following drug product infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Participants
  On or after Rel Day 60 | 14
  On or after Rel Day 100 | 7

20. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant Changes in Laboratory Parameters by Month 24
Description: Laboratory parameters included Hematology (Leukocytes [with a threshold range <4.0 x 10^9/L, >=18 x 10^9/L], Neutrophils [<1.0 x 10^9/L], Erythrocytes [<=3.0 x 10^12/L], Platelets [<=75 x 10^9/L]); Clinical chemistry (Sodium [<=126 millimoles per liter (mmol/L), >=156 mmol/L], Potassium [<=3 mmol/L, >=6 mmol/L], Glucose [<=3.0 mmol/L]), Renal (Urea Nitrogen [>=10.7 mmol/L], Creatinine [>=150 umol/L]) and liver (Alanine Aminotransferase [ALA]. Aspartate Aminotransferase [ASA], Alkaline Phosphatase [AP] with threshold range of >=3 x upper limit of normal (ULN), Bilirubin [>=34.2 micromoles per liter (umol/L)]). Clinical significance was decided by investigator.
Time Frame: From Day 1 to Month 24
Population: ITT population consisted of participants who initiated any study procedures, beginning with mobilization by G-CSF.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Percentage of participants
  Hematology: Leukocytes (<4.0 x 10^9/L) | 100.0
  Hematology: Leukocytes (>=18 x 10^9/L) | 2.9
  Hematology: Neutrophils (<1.0 x 10^9/L) | 97.1
  Hematology: Erythrocytes (<=3.0 x 10^12/L) | 71.4
  Hematology: Platelets (<=75 x 10^9/L) | 100.0
  Hematology: Hemoglobin (<=8.0 g/dL) | 77.1
  Liver: ALA (>=3 x ULN) | 11.4
  Liver: ASA (>=3 x ULN) | 5.7
  Liver: AP (>=3 x ULN) | 0.0
  Liver: Bilirubin (>=34.2 umol/L) | 0.0
  Renal: Urea Nitrogen (>=10.7 mmol/L) | 0.0
  Renal: Creatinine (>=150 umol/L) | 0.0
  Chemistry: Sodium (<=126 mmol/L) | 0.0
  Chemistry: Sodium (>=156 mmol/L) | 0.0
  Chemistry: Potassium (<=3 mmol/L) | 25.7
  Chemistry: Potassium (>=6 mmol/L) | 0.0
  Chemistry: Glucose (<=3.0 mmol/L) | 0.0

21. Secondary Outcome: Number of Emergency Room Visits (Post-Neutrophil Engraftment) by Month 24
Description: Number of emergency room visits (post-neutrophil engraftment) up to Month 24 were reported.
Time Frame: From Post-Neutrophil Engraftment up to Month 24
Population: Successful Neutrophil Engraftment Population (NEP) consisted of participants who achieved neutrophil engraftment defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion nadir) obtained on different days by Rel Day 43.
Measure: Number; unit: Emergency room visits
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Emergency room visits | 9

22. Secondary Outcome: Median Number of Emergency Room Visits (Post-Neutrophil Engraftment) by Month 24
Description: Median number of emergency room visits (post-neutrophil engraftment) up to Month 24 were reported.
Time Frame: From Post-Neutrophil Engraftment up to Month 24
Population: Successful NEP consisted of participants who achieved neutrophil engraftment defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion nadir) obtained on different days by Rel Day 43. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Median number of emergency room visits
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 9
Median number of emergency room visits | 1.0 [1 to 4]

23. Secondary Outcome: Number of In-patient Hospitalizations (Post-Neutrophil Engraftment) by Month 24
Description: Number of In-patient hospitalizations (post-neutrophil engraftment) by Month 24 were reported.
Time Frame: From Post-Neutrophil Engraftment up to Month 24
Population: Successful NEP consisted of participants who achieved neutrophil engraftment defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion nadir) obtained on different days by Rel Day 43.
Measure: Number; unit: Hospitalizations
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Hospitalizations | 17

24. Secondary Outcome: Median Number of In-patient Hospitalizations (Post-Neutrophil Engraftment) by Month 24
Description: Median number of In-patient hospitalizations (post-neutrophil engraftment) by Month 24 were reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: as for outcome 22
Measure: Median (Full Range); unit: Median number of hospitalization
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 17
Median number of hospitalization | 1.0 [1 to 4]

25. Secondary Outcome: Duration of In-patient Hospitalizations (Post-Neutrophil Engraftment) up to Month 24
Description: Duration of in-patient hospitalizations was calculated as: Duration = (Date of hospital discharge) - (Date of hospital admission before NE) + 1. Duration of In-patient hospitalizations (post-neutrophil engraftment) up to Month 24 was reported. The range of in-patient hospitalizations is influenced by hospital stays for participants who received allogeneic stem cell transplants.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: as for outcome 22
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 17
Days | 4.0 [2 to 56]

26. Secondary Outcome: Number of Intensive Care Units (ICU) Stays (Post-neutrophil Engraftment) by Month 24
Description: Number of ICU Stays (Post-neutrophil Engraftment) By Month 24 were reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: as for outcome 23
Measure: Number; unit: ICU Stays
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
ICU Stays | 0

27. Secondary Outcome: Duration of ICU Stays (Post-neutrophil Engraftment) by Month 24
Description: Duration of ICU Stays was calculated as: Duration = (Date of hospital discharge) - (Date of hospital admission before NE) + 1. Duration of ICU Stays (Post-neutrophil Engraftment) by Month 24 was reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: Successful NEP consisted of participants who achieved neutrophil engraftment defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion nadir) obtained on different days by Rel Day 43. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. No participant had ICU stay, hence data could not be estimated.
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 0

28. Secondary Outcome: Number of Participants Who Tested Positive and Negative for Vector-Derived Replication Competent Lentivirus (RCL) Detected by Month 24
Description: Number of participants who tested positive and negative for vector-derived RCL detected at Month 24 were reported. Screening of participant's blood samples for RCL at Month 24 following Lenti-D Drug infusion was performed, with the more rigorous co-culture assays used to distinguish any false positives as applicable.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Participants were evaluable if they have at least 1 RCL assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Participants
  Participants tested positive for RCL | 0
  Participants tested negative for RCL | 35

29. Secondary Outcome: Number of Participants With Insertional Oncogenesis by Month 24
Description: Insertional oncogenesis included myelodysplastic syndrome, leukemia, lymphoma. Number of participants with insertional oncogenesis at Month 24 were reported.
Time Frame: By Month 24 post-transplant
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 35
Participants | 1

ADVERSE EVENTS:
Time Frame: From date of informed consent up to Month 24
Arm/Group | Lenti-D Drug Product
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 22/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenti-D Drug Product (N=35)
Transaminases increased (Investigations) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 2 (2)
Visual field defect (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3)
Complication associated with device (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Aversion (Psychiatric disorders) | 1 (1)
Tic (Psychiatric disorders) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 2 (2)
Stenotrophomonas infection (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenti-D Drug Product (N=35)
Hypertension (Vascular disorders) | 8 (11)
Hypotension (Vascular disorders) | 3 (4)
Fatigue (General disorders) | 4 (6)
Pyrexia (General disorders) | 12 (20)
Catheter site pain (General disorders) | 17 (24)
Gait disturbance (General disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 3 (3)
Penile pain (Reproductive system and breast disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (17)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Agitation (Psychiatric disorders) | 6 (7)
Anxiety (Psychiatric disorders) | 3 (3)
Enuresis (Psychiatric disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 7 (14)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Blood creatinine increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (3)
International normalised ratio increased (Investigations) | 2 (2)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 3 (3)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 8 (12)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 8 (11)
Dizziness (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 14 (18)
Speech disorder (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 29 (44)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 (21)
Leukopenia (Blood and lymphatic system disorders) | 12 (19)
Lymphopenia (Blood and lymphatic system disorders) | 9 (13)
Neutropenia (Blood and lymphatic system disorders) | 29 (69)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 34 (54)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Dry eye (Eye disorders) | 5 (5)
Hypermetropia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 6 (6)
Visual impairment (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (21)
Abdominal pain upper (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 20 (31)
Dental caries (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 28 (60)
Stomatitis (Gastrointestinal disorders) | 34 (47)
Vomiting (Gastrointestinal disorders) | 26 (60)
Alopecia (Skin and subcutaneous tissue disorders) | 25 (29)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (9)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (4)
Haematuria (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 4 (5)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
BK virus infection (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 12 (14)
Device related infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 5 (5)
Human herpesvirus 6 infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 2 (2)
Otitis media acute (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (6)
Varicella (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 4 (7)
Pneumonia (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 22 (29)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03852498/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03852498/SAP_001.pdf